CLINICAL TRIAL: NCT06036693
Title: Mucopolysaccharidosis Patients in France in the Era of Specific Therapeutics
Brief Title: MPS (RaDiCo Cohort) (RaDiCo-MPS)
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C16-53
Record Dates: First submitted 2023-07-18; First posted 2023-09-14 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Mucopolysaccharidosis I; Mucopolysaccharidosis II; Mucopolysaccharidosis III; Mucopolysaccharidosis IV; Mucopolysaccharidosis VI; Mucopolysaccharidosis VII; Mucopolysaccharidosis IX; Multiple Sulfatase Deficiency Disease
MeSH Terms: conditions — Mucopolysaccharidosis I; Mucopolysaccharidosis II; Mucopolysaccharidosis III; Mucopolysaccharidosis IV; Mucopolysaccharidosis VI; Mucopolysaccharidosis VII; Multiple Sulfatase Deficiency Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to characterize the epidemiology and natural history of MPS diseases by building a retrospective and prospective collection of extensive phenotypic data from French MPS patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MPS based on clinically relevant enzyme deficiency, with abnormally elevated GAG urinary excretion and/or identification of pathogenic mutations.
* Signed informed consent or parents/guardian non-opposition for deceased patients (minor or protected major)

There are no non-inclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prevalent and incident patients will be included in the cohort RaDiCo-MPS.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-12-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the clinical data of MPS like growth for each system | Through study completion, an average of 5 years
Evaluation of the clinical data of MPS like signs for each system | Through study completion, an average of 5 years
Evaluation of the clinical data of MPS like symptoms for each system | Through study completion, an average of 5 years
Evaluation of the clinical data of MPS like complications for each system | Through study completion, an average of 5 years
Evaluation of the clinical data of MPS like psychomotor milestones | Through study completion, an average of 5 years
Evaluation of the clinical data of MPS like cognitive evolution | Through study completion, an average of 5 years
Evaluation of the clinical data of MPS like handicap using scales adapted to multivisceral disease for all types of MPS | Through study completion, an average of 5 years
Evaluation of the clinical data of MPS like handicap using scales adapted to cognitive and neurologic disease for the types I, II, III VII | Through study completion, an average of 5 years
Evaluation of the radiological data of MPS like standard bone radiographs | Through study completion, an average of 5 years
Evaluation of the radiological data of MPS like abdominal echography | Through study completion, an average of 5 years
Evaluation of the radiological data of MPS like echocardiography | Through study completion, an average of 5 years
Evaluation of the radiological data of MPS like cerebral and medullar tomodensitometry | Through study completion, an average of 5 years
Evaluation of the radiological data of MPS like magnetic resonance imaging | Through study completion, an average of 5 years
Evaluation of the electrophysiological data of MPS like EMG | Through study completion, an average of 5 years
Evaluation of the electrophysiological data of MPS like EEG | Through study completion, an average of 5 years
Evaluation of the electrophysiological data of MPS like ERG | Through study completion, an average of 5 years
Evaluation of the biochemical data of MPS like urinary GAG before specific treatment | Through study completion, an average of 5 years
Evaluation of the biochemical data of MPS like urinary GAG during specific treatment | Through study completion, an average of 5 years
Evaluation of the biochemical data of MPS like enzyme activities before specific treatment | Through study completion, an average of 5 years
Evaluation of the biochemical data of MPS like enzyme activities during specific treatment | Through study completion, an average of 5 years
Evaluation of the biochemical data of MPS like specific antibodies | Through study completion, an average of 5 years
Evaluation of the molecular data of MPS | Through study completion, an average of 5 years

SECONDARY OUTCOMES:
Description of the management of MPS diseases without specific treatment | Through study completion, an average of 5 years
Description of the management of MPS diseases before specific treatment | Through study completion, an average of 5 years
Description of the management of MPS diseases under specific treatment. | Through study completion, an average of 5 years
Description of the outcome of MPS diseases without specific treatment | Through study completion, an average of 5 years
Description of the outcome of MPS diseases before specific treatment | Through study completion, an average of 5 years
Description of the outcome of MPS diseases under specific treatment. | Through study completion, an average of 5 years
Identification of mutation(s) in each MPS type | Through study completion, an average of 5 years
Establishment of genotype/phenotype relationships in each MPS type. | Through study completion, an average of 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Thierry BILLETTE DE VILLEMEUR, Principal Investigator — INSERM UMR 1141
Locations (23):
- France (23):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Hôpital des Enfants - Groupe Hospitalier Pellegrin, Bordeaux
  - Hôpital Morvan, Brest
  - Hôpital d'Estaing, Clermont-Ferrand
  - Hôpital Beaujon, Clichy
  - Hôpital Raymond-Poincaré, Garches
  - Hôpital Jeanne de Flandre, Lille
  - Hôpital de la Timone, Marseille
  - Hôpital Gui de Chauliac, Montpellier
  - Hôpital Brabois, Nancy
  - Hôpital Armand Trousseau, Paris
  - Hôpital de la Croix Saint-Simon, Paris
  - Hôpital de la Pitié-Salpêtrière, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - Hôpital Robert Debré, Paris
  - Centre Hospitalier de Pau, Pau
  - American Memorial Hospital, Reims
  - Hôpital Pontchaillou, Rennes
  - Hôpital Charles Nicolle, Rouen
  - Hôpital de Hautepierre, Strasbourg
  - Clinique Monié, Toulouse
  - Hôpital des Enfants, Toulouse
  - Hôpital Clocheville, Tours